CLINICAL TRIAL: NCT01891994
Title: Extended Dosing With Eltrombopag in Refractory Severe Aplastic Anemia
Brief Title: Extended Dosing With Eltrombopag for Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130133; 13-H-0133; NCT01891994 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Cytokine; Hematopoiesis; Autoimmunity; Thrombocytopenia; Neutropenia
MeSH Terms: conditions — Anemia, Aplastic; Autoimmune Diseases; Thrombocytopenia; Neutropenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Administration of eltrombopag at a dose of 150mg/day for 6 months
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Oral administration of eltrombopag 150mg/day (75 mg/day for East Asian ancestry) for 6 months
  Other Names: Promacta

SUMMARY:
Background:

- Eltrombopag is a drug being tested for treating severe aplastic anemia. It can help improve blood counts in these patients. However, researchers do not know how long the drug can and should be taken for this type of anemia.

Objectives:

- To look at whether 6 months of treatment with eltrombopag can improve patient s blood counts.

Eligibility:

- Individuals at least 2 years of age who are taking eltrombopag for severe aplastic anemia.

Design:

* Participants will take eltrombopag by mouth once a day for 6 months.
* Blood samples will be collected every 2 weeks for the first 6 months. Bone marrow samples will be collected at 3 and 6 months. These samples will look at the effects of the study drug on the marrow.
* Participants will continue to take the study drug for as long as it is effective and if the side effects are not severe.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening blood disease that can be successfully treated with immunosuppressive drug regimens or allogeneic stem cell transplantation. However, 20-40% of patients are ineligible for transplant due to lack of an appropriate donor, age, or comorbidities. Immunosuppression can be more broadly utilized, but about 1/3 of patients do not respond to a single course of horse ATG and cyclosporine and have persistent severe cytopenias. Among patients who do respond to immunosuppression, responses may be partial, with persistent thrombocytopenia, neutropenia, and/or anemia. About 30% of responding patients either relapse or are dependent on continued cyclosporine administration. Patients with refractory severe cytopenias are at risk of dying from infection or bleeding, and they require regular platelet and/or red blood cell transfusions, which are expensive and inconvenient, Patients with refractory SAA are also at risk for progression to other hematologic disorders, including myelodysplasia and leukemia.

Thrombopoietin (TPO) was first identified as the principal protein regulating platelet production, and it stimulates the proliferation of megakaryocytes and release of platelets. TPO was later shown to stimulate proliferation of more primitive bone marrow stem and progenitor cells in vitro and in animal models, suggesting it could have an impact of production of red and white blood cells as well as platelets.

The 2nd generation oral small molecule TPO-agonist eltrombopag (Promacta ) has been shown to increase platelets in healthy subjects and in thrombocytopenic patients with chronic immune thrombocytopenic purpura (ITP) and hepatitis C virus (HCV)-infection. Eltrombopag has been well-tolerated in clinical trials, and unlike recombinant TPO, it does not induce autoantibodies. Eltrombopag received FDA accelerated approval on November 20, 2008 for the treatment of thrombocytopenia in patients with chronic immune (idiopathic) thrombocytopenic purpura who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy. In November 2012, FDA approval was received for hepatitis C associated thrombocytopenia.

We conducted a pilot dose finding study in patients with severe aplastic anemia who had refractory thrombocytopenia following standard immunosuppressive therapy. Patients began at a dose of 50 mg/day and escalated every two weeks to a maximum dose of 150 mg/day. We reported that 11 of 25 patients (44%) achieved hematological response in at least one lineage following 12 weeks of dose-escalating eltrombopag therapy, with minimal toxicity. Responding patients as assessed at 12 weeks were invited to continue on drug in an extension phase. With a median follow-up of 27 months on drug, 7 eventually became tri-lineage responders. Nine became transfusion-independent for platelets (median increase in platelet count 34,000/micro l), six had improved hemoglobin levels (median increase of 3.8g/dL), including three previously dependent on red cell transfusions achieving transfusion-independence, and eight exhibiting increased neutrophil counts (median increase 590 cells/mico L). Serial bone marrow biopsies demonstrated normalization of tri-lineage hematopoiesis in responders, without increased fibrosis.

In the previous study, response assessment occurred at 12 weeks, and patients not fulfilling response criteria at that time had the drug discontinued. Several patients began to have detectable changes in transfusion requirements or blood counts by 12 weeks, but did not fulfill response criteria by that time point and therefore had to discontinue eltrombopag. Other patients who barely met response criteria at 12 weeks showed very marked further improvements in blood counts in all lineages during the extension phase, in some cases not reaching maximal responses until one year after initiating eltrombopag. We hypothesize that a larger fraction of patients may respond if eltrombopag is continued for longer than 12 weeks.

We, therefore propose a follow-up Phase 2 study giving eltrombopag treatment for 24 weeks prior to definitive response assessment, and initiating study medication at a fixed dose of 150 mg/day (75 mg /day for individuals of East Asian ethnicity), given lack of toxicity at that dose in the prior study, and no evidence for response in any patient during dose escalation prior to reaching this dose. Responses will be assessed in all three lineages. Subjects with platelet, red cell, and/or neutrophil responses at 24 weeks may continue study medication (extended access) until they meet off study criteria.

The primary objective is to assess the efficacy of 6 months of eltrombopag administration in improving bone marrow function in SAA patients with persistent severe cytopenias refractory to treatment with immunosuppressive treatment.

Secondary objectives include assessment of relapse or clonal evolution, pre-treatment characteristics predicting response, and the impact of treatment and treatment response on quality of life.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Previous diagnosis of refractory severe aplastic anemia and following at least one treatment course of immunosuppression with a regimen containing antithymocyte globulin, alemtuzumab or cyclophosphamide.
* One or more of the following three clinically-significant cytopenias: platelet count less than or equal to 30,000/micro L or platelet-transfusion-dependence (requiring at least 4 platelet transfusions in the 8 weeks prior to study entry); neutrophil count less than 500/micro L; hemoglobin less than 9.0 g/dL or red cell transfusion-dependence (requiring at least 4 units of PRBCs in the eight weeks prior to study entry)
* Age greater than or equal to 2 years old
* Weight > 12 kg

EXCLUSION CRITERIA:

* Infection not adequately responding to appropriate therapy
* Evidence of a clonal disorder on cytogenetics performed within 12 weeks of study entry.
* Creatinine > 2.5 mg/dL
* Direct Bilirubin > 2.0 mg/dL
* SGOT or SGPT >5 times the upper limit of normal
* Hypersensitivity to eltrombopag or its components<TAB>
* Female subjects who are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
* Unable to understand the investigational nature of the study or give informed consent
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 7-10 days is likely
* Treatment with ATG, cyclophophamide or alemtuzamab within 6 months of study entry.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06-28; Primary Completion 2017-10-16 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E Dunbar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zhao Z, Sun Q, Sokoll LJ, Streiff M, Cheng Z, Grasmeder S, Townsley DM, Young NS, Dunbar CE, Winkler T. Eltrombopag mobilizes iron in patients with aplastic anemia. Blood. 2018 May 24;131(21):2399-2402. doi: 10.1182/blood-2018-01-826784. Epub 2018 Apr 9. No abstract available. PMID 29632023
- [Derived] Winkler T, Fan X, Cooper J, Desmond R, Young DJ, Townsley DM, Scheinberg P, Grasmeder S, Larochelle A, Desierto M, Valdez J, Lotter J, Wu C, Shalhoub RN, Calvo KR, Young NS, Dunbar CE. Treatment optimization and genomic outcomes in refractory severe aplastic anemia treated with eltrombopag. Blood. 2019 Jun 13;133(24):2575-2585. doi: 10.1182/blood.2019000478. Epub 2019 Apr 16. PMID 30992268
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0133.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag: Eltrombopag was administered for 6 months at a dose of 150mg daily in patients > 12 years of age, 75mg daily for patients 6 to 11 years of age, and 2.5 mg/kg/day for children 2-5 years of age. Dosing was reduced to 50% for patients of East Asian ethnicity.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag: Eltrombopag was administered for 6 months at a dose of 150mg daily in patients > 12 years of age, 75mg daily for patients 6 to 11 years of age, and 2.5 mg/kg/day for children 2-5 years of age.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 25
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 25
  More than one race | 4
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug Response as Defined by Clinically-signficant Hematologic Improvements
Description: Defined as unilineage or multilineage recovery by 1 or more of the following: 1) platelet response (increase to 20 × 103/μL above baseline or stable platelet counts with transfusion independence for a minimum of 8 weeks in those who were transfusion dependent on entry into the protocol); (2) erythroid response (when pretreatment hemoglobin was <9 g/dL, defined as an increase in hemoglobin by 1.5 g/dL or, in transfused patients, a reduction in the units of packed red blood cell transfusions by an absolute number of at least 4 transfusions for 8 consecutive weeks, compared with the pretreatment transfusion number in the previous 8 weeks); and (3) neutrophil response (when pretreatment absolute neutrophil count [ANC] of <0.5 × 103/μL as at least a 100% increase in ANC, or an ANC increase >0.5 × 103/μL, and the toxicity profile as measured using Common Terminology Criteria for Adverse Events).
Time Frame: 24 weeks
Population: All subjects who received Eltrombopag were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 40
Participants | 20

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 13/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=40)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Otitis media (Ear and labyrinth disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Infusion related reaction (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Urticaria (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=40)
Acute Myeloid Leukaemia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 16
Conjunctival pallor (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Ocular icterus (Blood and lymphatic system disorders) | 10
Petechiae (Blood and lymphatic system disorders) | 9
Purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Dizziness (Cardiac disorders) | 8
Dyspnoea (Cardiac disorders) | 8
Localised oedema (Cardiac disorders) | 1
Oedema peripheral (Cardiac disorders) | 9
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Syncope (Cardiac disorders) | 1
Ear Infection (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 3
External ear inflammation (Ear and labyrinth disorders) | 1
Otitis externa (Ear and labyrinth disorders) | 2
Otitis media (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Macular cyst (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 8
Anogenital warts (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 9
Dysgeusia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lip infection (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Oral candidiasis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Oropharyngeal pain (Gastrointestinal disorders) | 3
Pelvic pain (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Tooth infection (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 5
Decreased appetite (General disorders) | 5
Fatigue (General disorders) | 3
Flushing (General disorders) | 1
Hot flush (General disorders) | 3
Influenza like illness (General disorders) | 3
Infusion related reaction (General disorders) | 3
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 4
Mucosal infection (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Systemic inflammatory response syndrome (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic cyst (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 4
Psoriasis (Immune system disorders) | 1
Rhinitis allergic (Immune system disorders) | 2
Cellulitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 6
Soft tissue infection (Infections and infestations) | 1
Trichomoniasis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 5
Blister (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 8
Fracture (Injury, poisoning and procedural complications) | 2
Iron overload (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Computerised tomogram (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 5
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 6
White blood cell count decreased (Investigations) | 9
Dehydration (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Nonallopathic lesions of head region, not elsewhere classified (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 11
Insomnia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Urinary incontinence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Arteriosclerosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT01891994/Prot_SAP_000.pdf